CLINICAL TRIAL: NCT00680940
Title: Open Label, Randomized Multicentric Phase II Clinical Trial of Mycobacterium w in Combination With Paclitaxel Plus Cisplatin Versus Paclitaxel and Cisplatin in Advanced Non Small Cell Lung Cancer.
Brief Title: A Study of Mycobacterium w in Combination With Paclitaxel Plus Cisplatin in Advanced Non Small Cell Lung Cancer
Acronym: NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cadila Pharnmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-60/7260
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — TP protocol; Mycobacterium w vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy (Active Comparator): Paclitaxel + Cisplatin
  Interventions: Drug: Paclitaxel & Cisplatin
- Chemoimmunotherapy (Experimental): Paclitaxel + Cisplatin + Mycobacterium w
  Interventions: Biological: Mycobacterium w.

INTERVENTIONS:
Drug: Paclitaxel & Cisplatin — Chemotherapeutic agent
  Arms: Chemotherapy
Biological: Mycobacterium w. — Immunomodulator
  Arms: Chemoimmunotherapy

SUMMARY:
The purpose of this study is to determine whether Mycobacterium w in combination with Paclitaxel plus Cisplatin are effective in Advanced Non Small Cell Lung cancer.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) accounts for 75% of all lung cancers. majority of patients of NSCLC patients are stage IIIA or IIIB patients are suitable for radiotherapy, which could not improve the survival rates of 5-10%. This study proposed Mycobacterium w (heat killed) in combination chemotherapy of Cisplatin and Paclitaxel along with radiotherapy for adjuvant therapy management of NSCLC in controlled clinical trial, which may prove the efficacy, better survival rate and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Histologically or cytologically confirmed Non-Small Cell Cancer, Stage IIIB or IV.
* Age should be 18 years or above.
* ECOG should be in 0-1 range.
* Absolute neutrophil count ≥ 1,00,000/mm3
* hemoglobin ≥ 9.0g/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)range of institution (5times ULN if liver metastasis present).
* bilirubin not greater than 1.5 times ULN range of institution (3 times ULN if liver involvement).
* Creatinine ≤ upper limit of normal (ULN) range of institution.
* Negative pregnancy test for women of child bearing potential prior to entry into the trial.

Exclusion Criteria:

* Patient who have cytotoxic chemotherapy or radiotherapy prior to entering the study
* Patient with systematic brain metastasis.
* History of allergic reaction attributed to paclitaxel, cisplatin or mycobacterium w or any of their ingredients.
* Pregnant women or nursing women.
* Uncontrolled intercurrent illness that would limit compliance with study requirements.
* HIV positive patients.
* Previous splenectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Overall survival time of patients, quality of life | 12 months

SECONDARY OUTCOMES:
Response rate, Hematological toxicity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: R K Chaudhary, MD, Principal Investigator — Acharya Tulsi Regional Cancer Treatment & Research Institute; Rajeev Gupta, MD, Principal Investigator — Patel Hospital Pvt. Ltd.; Anup Majumdar, MD, Principal Investigator — Institute of Post Graduate Medical Education & Research; A. Rajkumar, MD, Principal Investigator — V.N. Cancer Center GKNM Hospital; Rajeev Seam, MD, Principal Investigator — Regional Cancer center, Indira Gandhi Medical College; A.K. Patel, MD, Principal Investigator — Choithram Hospital and Research Centre; Chanchal Goswami, MD, Principal Investigator — B.P.Poddar Hospital and Medical Research Ltd.; Jaydip Biswas, MD, Principal Investigator — Chittaranjan National Cancer Institute; Ritwik Pandyea, MD, Principal Investigator — Netaji Subhash Chandra Bose Cancer Research Institute; Aloke G Dastidar, MD, Principal Investigator — Bankura Sammilani Medical College; Narayanankutty Warrier, MD, Principal Investigator — Malabar Institute of Medical Science (MIMS); Ashutosh N Aggarwal, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Apurva Patel, MD, Principal Investigator — Gujarat Cancer & Research Institute; Santanu Chaudhary, MD, Principal Investigator — R.S.T. Cancer Hospital & Research Centre; Rajeev Prasad, MD, Principal Investigator — Regional Cancer Centre, Indira Ghandhi Institute of Medical Science; Ramakrishna Malladi, MD, Principal Investigator — MNJ Institute of Oncology, Regional Cancer Centre
Locations (14):
- India (14):
  - Gujarat Cancer & Research Institute, New Civil Hospital Campus, Asarwa, Ahmedabad
  - Regional Cancer Center, Indira Gandhi Medical College, Shimla, Himachal Pradesh
  - MNJ Institute of Oncology, Regional Cancer Centre, Red Hills, Hyderabad
  - Malabar Institute of Medical Science (MIMS), Calicut, Kerala
  - B.P. Poddar Hospital and Medical Research Ltd., New Alipore, Kolkata
  - Choithram Hospital and Research Centre, Indore, Madhya Pradesh
  - Regional Cancer Centre, Indira Gandhi Institute of Medical Science, Sheikhpura, Patna
  - Patel Hospital Pvt. Ltd, Jalandhar, Punjab
  - Acharya Tulsi Regional Cancer Treatment & Research Institute, Bikaner, Rajasthan
  - V.N. Cancer Center, GKNM Hospital, Coimbatore, Tamil Nadu
  - Netaji Subash Chandra Bose Cancer Research Institute, Kolkata, West Bangal
  - Bankura Sammilani Medical College, Gobindnagar, West Bengal
  - Institute of Post Graduate Medical education & Research, Kolkata, West Bengal
  - Chittaranjan National Cancer Institute, Kolkata, West Bengal